CLINICAL TRIAL: NCT00863291
Title: Phase 3 Study of the Effects of Buprenophine as Add-on Treatment to Antidepressants in Treating Acutely Suicidal Depressed Inpatients
Brief Title: A Double-Blind Study of Buprenorphine Treatment of Acute Suicidality
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abarbanel Mental Health Center (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HFDR-001-07
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Depression; Suicidal Ideation; Suicidal Action
Keywords: Depression; suicidality; buprenorphine
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): buprenorphine (range = 0.2-1.6 mg/day, starting dose = 0.2 mg/day, N = 20)
  Interventions: Drug: buprenorphine
- 2 (Placebo Comparator): Placebo given in a manner similar to he active comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: buprenorphine — buprenorphine (range = 0.2-1.6 mg/day, starting dose = 0.2 mg/day, N = 20)
  Other Names: Subotex
  Arms: 1
Drug: placebo — Placebo in a manner similar to the active comparator
  Arms: 2

SUMMARY:
The acutely suicidal patient presents a complex and dangerous clinical dilemma. Many suicidal patients receive antidepressant medications, but the onset of action of these medications is at least three weeks, and despite their established antidepressant effect, they have not shown a clear anti-suicidal benefit. Psychoanalysts hypothesized that depression (often leading to suicidality) shares important characteristics with the psychological sequellae of object loss and separation distress. Endogenous opioids (endorphines) have been implicated in mediating social bonding and separation distress in mammals. Anecdotal evidence and several clinical studies found the mixed opioid agonist-antagonist buprenorphine to be an effective antidepressant with a rapid onset of action. It is therefore hypothesized that buprenorphine may be a novel and quick-acting treatment for acute suicidality, especially in the context of depression. The proposed double-blind study will examine the effect of buprenorphine on acutely suicidal inpatients. Depression, suicidality, and overall functioning will be assessed before, during and after a two-week buprenorphine/placebo trial. A small subgroup of patients will also be treated with short-term psychoanalytic psychotherapy throughout the study period. It is hypothesized that subjects who receive the active drug will show rapid improvements in objective and subjective measures of suicidality and depression.

ELIGIBILITY:
Inclusion Criteria:

* depression

Exclusion Criteria:

* substance or alcohol abuse
* psychosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in suicidality as expressed by the score on the Beck Suicidal Ideation Scale | 2 weeks

SECONDARY OUTCOMES:
Reduction in psychache as measured by the OMMP | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Yovel, MD, PHD, Study Chair — Haifa University, Israel
Locations (1):
- Abarbanel MHC, Bat Yam, Israel

REFERENCES:
- [Background] Panksepp J. Neuroscience. Feeling the pain of social loss. Science. 2003 Oct 10;302(5643):237-9. doi: 10.1126/science.1091062. PMID 14551424